CLINICAL TRIAL: NCT06221137
Title: Laser Verses Conventional Circumferential Supracrestal Fiberotomy in Orthodontic Extrusion for Crown Lengthening: A Randomized Controlled Clinical Trial
Brief Title: Laser Verses Conventional Circumferential Supracrestal Fiberotomy in Orthodontic Extrusion for Crown Lengthening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, roquaiya eldardear, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7-12-22
Record Dates: First submitted 2023-07-11; First posted 2024-01-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Circumferential Supracrestal Fiberotomy; Orthodontic Extrusion; Crown Lengthening
Keywords: fiberotomy; extrusion; crown lengthening

STUDY DESIGN:
Intervention Model Description: Parallel groups, two arm, superiority Randomized Controlled Clinical Trial, with 1:1 allocation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional circumferential supracrestal fiberotomy (Active Comparator): * The amount of tooth that need to be extruded will be measured Bonding brackets slot 0,022"x0.028" Roth prescription on piggyback for the tooth with (0.016". x 0.022 ") stainless steel main arch wire and 0.0014" nickel titanium auxiliary.
    • Fiberotomy After 2 days of bonding, local anaesthetic solution will be administrated. The depth of the fibrotomy should be equal to the amount of tooth that need to be extruded.
  * supracrustal fibrotomy will be performed using 15 c blade (Carvalho, Bauer et al. 2006)
  Interventions: Procedure: conventional circumferential supracrestal fiberotomy
- laser circumferential supracrestal fiberotomy (Active Comparator): * The amount of tooth that need to be extruded will be measured
  * Bonding brackets slot 0,022"x0.028" Roth prescription
  * piggyback for the tooth with (0.016". x 0.022 ") stainless steel main arch wire and 0.0014" nickel titanium auxiliary.
    • Fiberotomy
  * After 2 days of bonding, local anaesthetic solution will be administrated.
  * The depth of the fibrotomy should be equal to the amount of tooth that need to be extruded.
  * A diode laser of 980 nm wavelength will be used The laser tip will be inserted, and incision will be extended around tooth circumference with the system configured to a continuous wave with the movement of the laser tip in an up and down stroking movement The laser tip will be moved in a circumferential manner taking care that all the fibers are lysed.
  Interventions: Procedure: laser circumferential supracrestal fiberotomy

INTERVENTIONS:
Procedure: conventional circumferential supracrestal fiberotomy — The amount of tooth that need to be extruded will be measured Bonding brackets slot 0,022"x0.028" Roth prescription on piggyback for the tooth with (0.016". x 0.022 ") stainless steel main arch wire and 0.0014" nickel titanium auxiliary.
  • Fiberotomy After 2 days of bonding, local anaesthetic solution will be administrated. The depth of the fibrotomy should be equal to the amount of tooth that need to be extruded.
  supracrustal fibrotomy will be performed using 15 c blade (Carvalho, Bauer et al. 2006)
  Arms: conventional circumferential supracrestal fiberotomy
Procedure: laser circumferential supracrestal fiberotomy — * The amount of tooth that need to be extruded will be measured
  * Bonding brackets slot 0,022"x0.028" Roth prescription
  * piggyback for the tooth with (0.016". x 0.022 ") stainless steel main arch wire and 0.0014" nickel titanium auxiliary.
    • Fiberotomy
  * After 2 days of bonding, local anaesthetic solution will be administrated.
  * The depth of the fibrotomy should be equal to the amount of tooth that need to be extruded.
  * A diode laser of 980 nm wavelength will be used The laser tip will be inserted, and incision will be extended around tooth circumference with the system configured to a continuous wave with the movement of the laser tip in an up and down stroking movement The laser tip will be moved in a circumferential manner taking care that all the fibers are lysed.
  Arms: laser circumferential supracrestal fiberotomy

SUMMARY:
The aim of this study is to the evaluate the stability of the amount of healthy tooth structure exposed after laser versus conventional technique of fiberotomy during orthodontic extrusion.

DETAILED DESCRIPTION:
Parallel groups, two arm, superiority Randomized Controlled Clinical Trial, with 1:1 allocation.

PICO:

Population: patients with endodontically treated teeth and short clinical crown that require crown lengthening in the esthetic zone Intervention: laser fiberotomy with orthodontic extrusion Control: conventional fiberotomy using blade with orthodontic extrusion

Outcomes:

Primary outcome: Stability of the mount of healthy tooth structure exposed.

Secondary outcomes:

* Stability of gingival Margin reference.
* Stability of the alveolar bone.
* Rate of tooth extrusion.
* Sulcus depth.
* Pain Time: 8 weeks after retention

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* Teeth in the esthetic zone
* Restorable teeth with successful endodontic treatment
* Adjacent teeth with clinical attachment of at least two-thirds of the root length, thus permitting adequate support for orthodontic movement
* Crown root ratio after extrusion of the needed ferrule amount not less than 1:1

Exclusion Criteria:

* Patients with bad oral hygiene or Periodontally affected teeth
* Uncontrolled diabetic patients
* Pregnant females
* Medications that could affect tooth movement (bisphosphonate) radiation therapy less than 2 years
* Moderate-to-heavy daily smokers (who report consuming at least 11 cigarettes/day)
* Teeth with periapical inflammation, ankylosis or vertical root fracture
* Teeth with probability of furcation exposure after extrusion.
* The level of the root is 3 mm or more apical to the level of the bone

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Stability of amount of healthy tooth structure exposed | 8 weeks after retention.
  Amount of healthy tooth structure exposed:
  This is measured from the 6 guide marks in the acrylic stent around the extruded teeth to the healthy tooth structure using UNC periodontal probe in millimeters.

SECONDARY OUTCOMES:
Stability of gingival Margin | 8 weeks after retention.
  This is measured from the 6 guide marks in the acrylic stent around the extruded teeth to the gingival margin using UNC periodontal probe in millimeters.
Stability of the alveolar bone | 8 weeks after retention.
  This is measured from the 6 guide marks in the acrylic stent around the extruded teeth to the top of the alveolar crest using UNC periodontal probe in millimeters.
  This is done after administration of local anesthesia by infiltration around the tooth
Rate of tooth extrusion | 8 weeks after retention.
  This is measured by calculating the average tooth extrusion per week by dividing the amount of healthy tooth structure exposed on the number of weeks.
Sulcus depth | 8 weeks after retention.
  The distance from gingival margin to the base of the sulcus in millimetres.
Post operative pain | 8 weeks after retention.
  VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Nesma M Shemais, PhD, Study Director — Cairo University; Heba A Akl, PhD, Study Director — Cairo University
Locations (1):
- focality of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No